CLINICAL TRIAL: NCT02340754
Title: Mindfulness-based Stress Reduction for Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Angela Senders, ND, MCR, Assistant Professor, National University of Natural Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MBSR-MS-001; 1K23AT008211-01A1 (NIH)
Record Dates: First submitted 2015-01-11; First posted 2015-01-19 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
Keywords: mindfulness; meditation; stress, psychological; quality of life; randomized controlled trial
MeSH Terms: conditions — Multiple Sclerosis; Stress, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness-base Stress Reduction (Experimental): Mindfulness-based stress reduction is a formalized, experiential, 8-week stress-management program. Participants attend weekly two-hour classes and a half-day retreat during which they learn mindfulness meditation, breath work, yoga postures, self-reflection and awareness.
  Interventions: Behavioral: Mindfulness-based Stress Reduction
- MS Education Control (Active Comparator): The MS Education Control program is matched to MBSR for time and attention yet has no overlap with intervention content. Each two-hour class uses a pamphlet published by the National MS Society to present information about a different MS topic such as Fatigue; Bowel and Bladder Problems; Diet; Spasticity; and Nutritional Supplementation: Vitamins, Minerals, and Herbs.
  Interventions: Behavioral: MS Education Control

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction
  Other Names: MBSR
  Arms: Mindfulness-base Stress Reduction
Behavioral: MS Education Control
  Arms: MS Education Control

SUMMARY:
The primary purpose of this study is to assess the feasibility of mindfulness-based stress reduction (MBSR) for adults with any type of multiple sclerosis. The secondary objectives are to: 1) Explore the ability of MBSR to improve perceived stress and quality of life compared to an education control group; and 2) Explore the durability of the effects of MBSR over one year.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or older
* Definite relapsing remitting, secondary progressive, or primary progressive MS by revised McDonald criteria;
* Expanded Disability Severity Scale ≤ 8 at baseline;
* Stable on MS disease modifying, anxiolytic, or antidepressant medications for three months prior to baseline visit;
* Mild to moderate stress defined by a score of ≥ 10 on the Perceived Stress Scale at screening;
* Ability to read and write in English;
* Willingness to provide informed consent and comply with study activities, including weekly MBSR sessions and daily practice or weekly Education Control classes.

Exclusion Criteria:

* MBSR or cognitive behavioral therapy training within the last 5 years;
* Current regular meditation or yoga practice (weekly or more often);
* MS exacerbation within 30 days of Baseline Visit;
* Mini-Mental Status Examination (MMSE) score of ≤ 26 at Screening Visit;
* Active suicidal ideation (Beck Depression Inventory) at Screening Visit;
* Reported or medically recorded diagnoses of current serious psychological disorders other than depression and anxiety;
* Other current life-threatening or severely disabling physical disorders;
* Positive pregnancy urine test at Baseline and women planning pregnancy during the study period (contraception not required);
* Cancer, other than basal or squamous skin cancers; or
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Recruitment: Number of participants enrolled over a ten-month period | Recruitment will be tracked monthly with an expected recruitment period of 10 months..
  Feasible recruitment is defined as the ability to recruit and enroll 60 participants with multiple sclerosis (MS) over a ten-month time frame. Recruitment rate will be calculated as the proportion of eligible patients who provided informed consent per month.
Adherence to Mindfulness-based Stress Reduction (MBSR): Number of Participants who are present for at least 5 of the classes, including the final class, and complete at least 70% of homework. | Baseline to 8 weeks
  Adherence will be tracked with a sign-in/sign out sheet at each class and with daily homework logs. Attendance will be calculated by a sign in/sign out sheet, being present for at least 75% of a class will count as attended. Homework will be tabulated as both a frequency count (number of days homework was completed) and amount (total number of minutes completed). Participants who are present for at least 5 of the classes, including the final class, and complete at least 70% of homework will be recorded as 'adherent'.
Adoption: Qualitative assessment of facilitators of and barriers to participation in the MBSR program. | Week 4 and week 8 of the 8 week intervention.
  Adoption is defined as the ability of participants to take part in activities such as yoga poses and meditative exercises. Qualitative outcomes include a brief, semi-structured focus group conducted at the beginning of the MBSR classes during weeks five and eight. Focus groups will address successes and any challenges participants may be experiencing. Focus groups will be audio recorded and transcribed verbatim for qualitative analysis.
Completion: Number of participants with complete follow-up at 12 months post-intervention. | 14 months
  A feasible completion rate is defined as complete follow-up in at least 70% of enrolled subjects at 12-months post-intervention. Completion indicates acceptability of a long-term trial and will inform future study designs.

SECONDARY OUTCOMES:
Change from baseline in Perceived Stress Scale at 8 weeks | Baseline and 8 weeks
Change in Perceived Stress Scale from 8 weeks to 12 months | 8 weeks and 12 months
Change from baseline in Short Form-36 Mental Health Subscale to 8 weeks | Baseline and 8 weeks
  Mental health-related quality of life.
Change in Short Form-36 Mental Health Subscale from 8 weeks to 12 months | 8 weeks and 12 months
  Mental health-related quality of life.
Change in baseline Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Score to 8 weeks | Baseline and 8 weeks
  PROMIS Computerized Adaptive Test of Anxiety
Change in PROMIS Anxiety Score from 8 weeks to 12 months | 8 weeks and 12 months
  PROMIS Computerized Adaptive Test of Anxiety
Change in baseline PROMIS Depression Score to 8 weeks | Baseline and 8 weeks
  PROMIS Computerized Adaptive Test of Depression
Change in PROMIS Depression Score from 8 weeks to 12 months | 8 weeks and 12 months
  PROMIS Computerized Adaptive Test of Depression
Change in baseline PROMIS Fatigue Score to 8 weeks | Baseline and 8 weeks
  PROMIS Computerized Adaptive Test of Fatigue
Change in PROMIS Fatigue Score from 8 weeks to 12 months | 8 weeks and 12 months
  PROMIS Computerized Adaptive Test of Fatigue
Change in baseline PROMIS Pain Score to 8 weeks | Baseline and 8 weeks
  PROMIS Computerized Adaptive Test of Pain
Change in PROMIS Pain Score from 8 weeks to 12 months | 8 weeks and 12 months
  PROMIS Computerized Adaptive Test of Pain

CONTACTS AND LOCATIONS:
Locations (1):
- National College of Natural Medicine, Portland, Oregon, United States

REFERENCES:
- [Background] Senders A, Bourdette D, Hanes D, Yadav V, Shinto L. Perceived stress in multiple sclerosis: the potential role of mindfulness in health and well-being. J Evid Based Complementary Altern Med. 2014 Apr;19(2):104-11. doi: 10.1177/2156587214523291. Epub 2014 Feb 20. PMID 24647090
- [Background] Senders A, Sando K, Wahbeh H, Peterson Hiller A, Shinto L. Managing psychological stress in the multiple sclerosis medical visit: Patient perspectives and unmet needs. J Health Psychol. 2016 Aug;21(8):1676-87. doi: 10.1177/1359105314562084. Epub 2014 Dec 19. PMID 25527612